CLINICAL TRIAL: NCT02831946
Title: Intracuticular Sutures Versus Glue (Dermabond) for Skin Closure After Cesarean Delivery
Brief Title: Suture Versus Glue (Dermabond) Closure During Cesarean Delivery
Acronym: SVGCS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yair Daykan, MD, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0062-16-MMC
Record Dates: First submitted 2016-06-14; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Adhesive; Band; Suture; Complications
Keywords: skin closure; intracuticular suture; glue (dermabond)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MODIFIED VICRYL PLUS (Experimental): The intra-cuticular layer will closed with with VICRYL PLUS suture
  Interventions: Device: MODIFIED VICRYL PLUS
- DERMABOND GLUE (Experimental): The intra-cuticular layer will closed with with DERMABOND GLUE
  Interventions: Device: DERMABOND GLUE

INTERVENTIONS:
Device: MODIFIED VICRYL PLUS — closing the intra-cuticular layer with MODIFIED VICRYL PLUS suture
  Arms: MODIFIED VICRYL PLUS
Device: DERMABOND GLUE — closing the intra-cuticular layer with Dermabond glue
  Arms: DERMABOND GLUE

SUMMARY:
To investigate the effect of intracutaneous suture closure versus Glue (dermabond) closure at cesarean section (CS) on long-term cosmetic and maternal outcome.

DETAILED DESCRIPTION:
Women undergoing planned CS were randomized to either intracutaneous suture closure or glue closure using a 1:1 allocation algorithm. Participants and outcome assessors were blinded to group allocation. Scar evaluation was performed after two months.

Primary outcome measures were Patient and Observer Scar Assessment Scale (POSAS) summary scores 2 months after surgery. Secondary outcome measures were, duration of surgery, and development of hematoma, seroma, surgical site infection (SSI) or wound disruption.

Data were analyzed according to the intention to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18 and 45 years
* Elective cesarian section

Exclusion Criteria:

* Clinical signs of infection at the time of CS
* History of keloids and a medical disorder that could affect wound healing
* Hypersensitivity to any of the suture materials used in the protocol
* Diabetes mellitus
* Disorders requiring chronic corticosteroid use or immunosuppression

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | 2 month
  Subjective scar rating will be performed using the patient component of the POSAS. The POSAS Scale consists of 2 numerical numeric scales: The Patient Scar Assessment Scale and the Observer Scar Assessment Scale

SECONDARY OUTCOMES:
post operative complication | 1 month
  Development of surgical site infection or wound disruption.

CONTACTS AND LOCATIONS:
Overall Officials: Reut Ohana, Principal Investigator — Meir Helsinki
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
within 6 m of finishing the study